CLINICAL TRIAL: NCT00872248
Title: Correlation of Neuraxial Anesthesia and Restless Leg Syndromes in Cesarean Delivery
Brief Title: Neuraxial Anesthesia and Restless Leg Syndromes in Cesarean
Acronym: NARELESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanjing Medical University (Other)
Responsible Party: XiaoFeng Shen, Nanjing Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NMU-200903-MZ005; NJFY09102M112
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-05

CONDITIONS: Cesarean Section; Restless Leg Syndrome
Keywords: Restless leg syndrome; Spinal anesthesia; Epidural anesthesia; Neuraxial block
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Anesthesia, Spinal; Anesthesia, Epidural

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Parturients received spinal anesthesia
  Interventions: Procedure: Spinal anesthesia
- 2 (Active Comparator): Parturients received epidural anesthesia
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Spinal anesthesia — Procedures of spinal anesthesia with bupivacaine 0.5%, 10-15mg
  Other Names: Intrathecal anesthesia
  Arms: 1
Procedure: Epidural anesthesia — Procedures of epidural anesthesia with ropivacaine 0.75%, 75-120mg
  Other Names: Extradural anesthesia
  Arms: 2

SUMMARY:
The restless leg syndromes is a common sensorimotor disorder of unknown cause affecting approximately 10% of the population. Different literature had different views on the association between neuraxial anesthesia and the occurrence of restless leg syndrome. Some reported that spinal anesthesia induced postoperative restless leg syndrome, but other studies showed that spinal and general anesthesia all two did not cause restless leg syndrome. A potential difference amongst these studies is that a big difference exists in surgical types. The investigators proposed that different types of surgery performed undergoing various anesthesia, and that there is a big difference in original pathophysiological condition. Therefore, the investigators hypothesized that pregnant women who have special physical states would have had an association between neuraxial anesthesia and restless leg syndrome in such patients who received selective cesarean section undergoing spinal or epidural anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Healthy pregnancy
* Selective cesarean
* Gestational age >= 37 weeks
* Chinese

Exclusion Criteria:

* Allergic to local anesthetics
* Allergic to opioids
* History of psychosis
* Cognition malfunction
* Any organic diseases
* Original lower extremity dyskinesia and paraesthesia
* Chronic pain
* Difficult in sleep
* Drug and alcohol abuse

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2009-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Occurrence of restless leg syndrome | One day to one week after completion of cesarean

SECONDARY OUTCOMES:
Intraoperative anesthetic effectiveness | From the beginning of anesthesia (0 min) to completion of cesarean (45 min)
  The anesthetic efficacy of neuraxial anesthesia will be assessed with sensony and movement block means
Postoperative analgesic effectiveness | From the initiation of analgesia (0 min) to 48 h after cesarean
  This will be assessed with visual analog scale (VAS) of pain in a 0 to 10cm scoring bar
Other postoperative side effects: hypotension, pruritus, nausea, vomiting, distal paraesthesia, dyskinesia in lower extremity | From the completion of cesarean (1 day) to one week follow-up
Psychological state | From one day to one week follow-up after cesarean
  This will be assessed with self anxiety and depression scales
Infant weight | Three min after cesarean section
One-min Apgar score | One min after cesarean section
Five-min Apgar score | Five min after cesarean section
Intraoperative vital signs | From the beginning of cesarean (0 min) to completion of operation (45 min)

CONTACTS AND LOCATIONS:
Overall Officials: XiaoFeng Shen, MD, Study Director — Nanjing Medical University
Locations (1):
- Nanjing Maternal and Child Health Care Hospital, Nanjing, Jiangsu, China